CLINICAL TRIAL: NCT03965949
Title: Impact of Different Strategies in Frozen Cycles Using HRT in Normo Responding Patients Undergoing IVF/ICSI Cycles: a Multicenter Cohort Study
Brief Title: Different Strategies in Frozen IVF/ICSI Cycles
Status: Completed | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Siristatidis Charalampos, MD, PhD, Associate Professor in Obstetrics Gynaecology, National and Kapodistrian University of Athens
Other Study IDs: HRT001
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Pregnancy Rates

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Natural cycle, spontaneous ovulation or ovulation triggering by exogenous hCG without luteal support
  Interventions: Drug: Hormone Replacement cycle 1
- Group 2: Natural cycle, spontaneous ovulation or ovulation triggering by exogenous hCG with luteal support (progesterone)
  Interventions: Drug: Hormone Replacement cycle 1
- Group 3: Hormone Replacement cycle (cyclacur) plus GnRHa suppression with luteal support (progesterone)
  Interventions: Drug: Hormone Replacement cycle 2
- Group 4: Hormone Replacement cycle (cyclacur) without GnRHa suppression with luteal support (progesterone)
  Interventions: Drug: Hormone Replacement cycle 2

INTERVENTIONS:
Drug: Hormone Replacement cycle 1 — Hormone Replacement cycle (cyclacur) without GnRHa suppression with luteal support (progesterone)
  Groups: Group 1; Group 2
Drug: Hormone Replacement cycle 2 — Hormone Replacement cycle with GnRHa suppression
  Groups: Group 3; Group 4

SUMMARY:
In the absence of robust contemporary data, investigators decided to perform a multicenter cohort study of various IVF centers, to compare the different modalities used for pregnancy rates following frozen-thawed embryo transfer (FET) treatment cycles in normoovulatory patients undergoing IVF/ICSI.

DETAILED DESCRIPTION:
In general, the type of FET protocol for each patient is selected by the attending physicians at their own discretion. In all centers, patients with ovulatory cycles are typically prescribed an NC-FET or mNC-FET, whereas patients with oligomenorrhoea or amenorrhoea are prescribed an artificial cycle to prepare the endometrium for FET.

Ovarian stimulation protocol

1. The antagonist protocol
2. The long 21 /2 agonist protocol Laboratory technique

a. IVF or b. ICSI Embryo freezing using only vitrification will be performed in days 3 or 5/6. Embryo transfer will be conducted at days 3 or 5/6. The maximum number of embryos transferred will be two, as in accordance to the Hellenic legislation.

The following modalities will be analyzed, patients with:

1. Natural cycle, spontaneous ovulation or ovulation triggering by exogenous hCG without luteal support (Group 1)
2. Natural cycle, spontaneous ovulation or ovulation triggering by exogenous hCG with luteal support (progesterone) (Group 2)
3. Hormone Replacement cycle (cyclacur) plus GnRHa suppression with luteal support (progesterone) (Group 3)
4. Hormone Replacement cycle (cyclacur) without GnRHa suppression with luteal support (progesterone) (Group 4)

Of note, the conversion between different supplementation methods may be testimated as follows: 0.75 mg of micronised estradiol (oral administration) = 1.25 g of estradiol gel (transdermal administration) = 1 mg of estradiol valerate (oral or vaginal adminstration).

ELIGIBILITY:
Inclusion Criteria:

age 25-39 years, BMI ≤ 35 and ≥ 19, normo-ovulatory patients and basal FSH ≤11 mIU/mL. Definition of expected normal ovarian response will be based primarily on antral follicle count (AFC) between 6-14.

Exclusion Criteria:

history of more than three previous unsuccessful IVF/ICSI cycles, FSH > 12 mIU/mL, BMI >35 or <19, poor ovarian response according to the 2011 Bologna criteria, PCOS patients according to the Rotterdam criteria, history of untreated autoimmune, endocrine or metabolic disorders, history of pathology affecting the endometrial cavity and/or receptivity and clinical and/or laboratory markers of hereditary or acquired thrombophilia that complied to the standard protocols of each Unit and patients without embryo after thawing.

Ages: 25 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Following clinical evaluation along with previous medical and reproductive history, participants will be categorized according to the subfertility factor and further demographic parameters (age, Body Mass Index (BMI), smoking status, basal FSH levels, parity, antral follicle count (AFC) in the fresh cycle, type (primary/secondary) and duration of subfertility and number of unsuccessful IVF/ICSI attempts (fresh and/or frozen) will be recorded along with the respective hormonal profiles.
Sampling Method: Probability Sample
Enrollment: 311 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
live birth | 1 year
  birth after 20 weeks of gestation
ongoing pregnancy | 3 months
  positive heart rate after 12 weeks
miscarriage | 6 months
  pregnancy loss up to 20 weeks of gestation

SECONDARY OUTCOMES:
biochemical pregnancy (positive β-hCG), multiple, ectopic and clinical pregnancy rates | 3 months
  positive β-hCG, multiple, ectopic and clinical pregnancy rates

CONTACTS AND LOCATIONS:
Locations (1):
- Attikon University Hospital, Athens, Chaidari, Greece

IPD SHARING:
Plan to Share IPD: Undecided
Will discuss it with other authors